CLINICAL TRIAL: NCT07328178
Title: Analysis of the Role of IgE Proteoforms in Health and Disease
Acronym: IgE-PhD
Status: Recruiting | Type: Observational
Sponsor: KU Leuven (Other)
Responsible Party: Principal Investigator, Rik Schrijvers, Prof. Dr. Rik Schrijvers, Universitaire Ziekenhuizen KU Leuven
Other Study IDs: S69940
Record Dates: First submitted 2025-12-26; First posted 2026-01-09 (Actual); Last update posted 2026-01-09 (Actual); Status verified 2025-11

CONDITIONS: Anaphylaxis; Mastocytosis; X-linked Agammaglobulinaemia; Venom Allergy; Chronic Spontaneous Urticaria (CSU); Type I Allergy; Medication Allergy; Healthy Control; Hereditary Alpha-Tryptasemia
MeSH Terms: conditions — Anaphylaxis; Mastocytosis; Bruton type agammaglobulinemia; Venom Hypersensitivity; Chronic Urticaria; Drug Hypersensitivity; Hereditary alpha-tryptasemia syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (9):
- Healthy controls
  Interventions: Other: Blood sample collection
- Patients with type I allergy: Including medication allergy, venom allergy, food allergy, allergic rhinitis
  Interventions: Other: Blood sample collection
- Patients with chronic spontaneous urticaria: With or without omalizumab
  Interventions: Other: Blood sample collection
- Patients with a recent history of anaphylaxis: In whom serial sampling can be performed
  Interventions: Other: Blood sample collection
- Patients undergoing desensitization for venom allergy
  Interventions: Other: Blood sample collection
- Patients undergoing desensitization for medication allergy
  Interventions: Other: Blood sample collection
- Patients with mastocytosis
  Interventions: Other: Blood sample collection
- Patients with hereditary alpha tryptasemia
  Interventions: Other: Blood sample collection
- Patients with X-linked agammaglobulinemia (XLA)
  Interventions: Other: Blood sample collection

INTERVENTIONS:
Other: Blood sample collection — Blood sample collection

SUMMARY:
The goal of this observational study is to evaluate the role of IgE proteoforms in healthy volunteers and in patients with type I allergy, patients with chronic spontaneous urticaria, patients with a recent history of anaphylaxis, patients with mastocytosis, patients with hereditary alpha tryptasemia, patients with X-linked agammaglobulinemia (XLA), and patients undergoing desensitization for venom or medication allergy.

ELIGIBILITY:
Inclusion Criteria:

* CSU and type I allergic diseases (including anaphylaxis and desensitization), atopic dermatitis, mastocytosis, XLA and HaT (informed consent, age: any available adult subject, gender: any available subject, clinical phenotype and specific information about the allergy (e.g. severity, medication, medical history, laboratory testing)
* Healthy controls (informed consent, age matched to the allergic patients, gender matched to the allergic patients, patient-reported symptoms related to allergy to aeroallergens, food, drugs, hymenoptera venom, CSU)

Exclusion Criteria:

* Absence of informed consent
* Age < 18 years old

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients with type I allergy (including medication allergy, venom allergy, food allergy, allergic rhinitis), patients with chronic spontaneous urticaria (with or without omalizumab), patients with a recent history of anaphylaxis in whom serial sampling can be performed, patients undergoing desensitization for venom allergy, patients undergoing desensitization for medication allergy, patients with mastocytosis, patients with hereditary alpha tryptasemia, patients with X-linked agammaglobulinemia (XLA), healthy controls
Sampling Method: Non-Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2025-01-01 (Actual); Primary Completion 2029-01-01 (Estimated); Study Completion 2029-01-01 (Estimated)

PRIMARY OUTCOMES:
Evaluation of IgE proteoforms | 4 years

CONTACTS AND LOCATIONS:
Overall Officials: Rik Schrijvers, MD, PhD, Principal Investigator — UZ/KU Leuven
Locations (1):
- UZ/KU Leuven, Leuven, Vlaams-Brabant, Belgium

IPD SHARING:
Plan to Share IPD: No